CLINICAL TRIAL: NCT02320526
Title: Interval-training in Type 2 Diabetics - Mechanisms Behind Increased Glucose Disposal and Effects on Systemic Inflammation
Brief Title: Interval-training in Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-6-2014-043
Record Dates: First submitted 2014-12-08; First posted 2014-12-19 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Training; Interval training; Systemic inflammation; Glucose disposal; Insulin sensitivity; Glucose effectiveness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Control intervention: Subjects will continue their life unaltered during the 14 days intervention period
  Interventions: Behavioral: Control
- Continuous walking (Experimental): Training intervention: Subjects will perform continuous walking for one hour per day at every weekday during the 14 days intervention period
  Interventions: Behavioral: Continuous walking
- Interval Walking (Experimental): Training intervention: Subjects will perform interval walking for one hour per day at every weekday during the 14 days intervention period. Interval walking will be performed as repeated cycles of three minutes of slow and hree minutes of fast walking during the entire training session
  Interventions: Behavioral: Interval walking

INTERVENTIONS:
Behavioral: Control
  Other Names: CON
  Arms: Control
Behavioral: Continuous walking
  Other Names: CWT
  Arms: Continuous walking
Behavioral: Interval walking
  Other Names: IWT
  Arms: Interval Walking

SUMMARY:
Interval training is superior to continuous training for improving glycemic control, hereunder glycemic variability and -spikes. However, the underlying mechanisms and the clinical impact is at present unknown.

The overall objective of this project is to determine the mechanisms underlying aeroic interval-training-induced reductions in glycemic variability and -spikes, and the impact on levels of systemic inflammation in type 2 diabetes patients. It is hypothesized that aerobic interval training reduces glycemic variability and -spikes more than continuous training due to larger improvements in both peripheral insulin sensitivity and the mass action effect of glucose. Moreover, it is hypothesized that these reductions in glycemic variability and -spikes also reduces systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* BMI >18 but <40 kg/m2

Exclusion Criteria:

* Pregnancy
* Smoking
* Contraindication to increased levels of physical activity
* More than moderate levels of physical activity (>90 min/week) of maximally moderate intensity
* Insulin dependence
* Thyroid, liver, lung, heart or kidney disease, with the need for treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Change from baseline at 14 days
  Glycemic control incl. glycemic variability and -spikes, will be measured with continuous glucose monitoring over 24 hours during standardized dietary intake before and after each intervention.

SECONDARY OUTCOMES:
Urinary isoprostanes as a measure of systemic inflammation | Change from baseline at 14 days
  Systemic inflammation will be measured as isoprostanes in urine collected over 24 hours. The changes in glycemic control (Outcome 1), will be correlated with the changes in systemic inflammation.
Rate of dissappearance during a 2-step (pancreatic + hyperinsulinemic) hyperglycemic clamp, as a measure of glucose effectiveness + insulin sensitivity | Change from baseline at 14 days
  A 2-step (pancreatic + hyperinsulinemic) hyperglycemic clamp will be performed before and after each intervention, to assess the mechanisms behind the intervention-induced improvements in glycemic control. In this way, the intervention-induced effects on glucose effectiveness and insulin sensitivity will be assessed.

OTHER OUTCOMES:
Resting energy expenditure and respiratory exchange rate | Change from baseline at 14 days
  Resting indirect calorimetry measurements will be performed before and after each intervention, to assess the effects of the interventions on resting energy-expenditure and respiratory exchange rates.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, PhD, Principal Investigator — Rigshospitalet, The Centre for Physical Activity Research
Locations (1):
- The Centre for Physical Activity Research, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Karstoft K, Clark MA, Jakobsen I, Knudsen SH, van Hall G, Pedersen BK, Solomon TPJ. Glucose effectiveness, but not insulin sensitivity, is improved after short-term interval training in individuals with type 2 diabetes mellitus: a controlled, randomised, crossover trial. Diabetologia. 2017 Dec;60(12):2432-2442. doi: 10.1007/s00125-017-4406-0. Epub 2017 Aug 25. PMID 28842722
- [Derived] Karstoft K, Brinklov CF, Thorsen IK, Nielsen JS, Ried-Larsen M. Resting Metabolic Rate Does Not Change in Response to Different Types of Training in Subjects with Type 2 Diabetes. Front Endocrinol (Lausanne). 2017 Jun 13;8:132. doi: 10.3389/fendo.2017.00132. eCollection 2017. PMID 28659869
- [Derived] Karstoft K, Clark MA, Jakobsen I, Muller IA, Pedersen BK, Solomon TP, Ried-Larsen M. The effects of 2 weeks of interval vs continuous walking training on glycaemic control and whole-body oxidative stress in individuals with type 2 diabetes: a controlled, randomised, crossover trial. Diabetologia. 2017 Mar;60(3):508-517. doi: 10.1007/s00125-016-4170-6. Epub 2016 Dec 9. PMID 27942800